CLINICAL TRIAL: NCT02648126
Title: Research of Pure Red Cell Aplasia in Patients With Chronic Kidney Disease and in Use of Epoetin Alfa Produced by Immunobiological Technology Institute (Bio-Manguinhos) From Oswaldo Cruz Foundation (Bio-Manguinhos / Fiocruz)
Brief Title: Pure Red Cell Aplasia in Patients With Chronic Kidney Disease and in Use of Epoetin Alfa
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ASCLIN 004/2014
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Red-Cell Aplasia, Pure; Renal Insufficiency, Chronic
MeSH Terms: conditions — Red-Cell Aplasia, Pure; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pure red cell aplasia participants (Other): Group of participants with pure red cell aplasia and chronic kidney disease, that have resistance criteria to treatment with epoetin alfa produced by Bio-Manguinhos / Fiocruz. The Patients who meet the appropriate criteria in the selection period will be subject to Pure Red Cell Aplasia diagnostic confirmation.
  Interventions: Procedure: Pure Red Cell Aplasia diagnostic confirmation

INTERVENTIONS:
Procedure: Pure Red Cell Aplasia diagnostic confirmation — Patients who meet the appropriate criteria in the selection period will be subject to Pure Red Cell Aplasia diagnostic confirmation by collecting 20 mL of blood in dialysis units.
  The samples will be processed, aliquoted and transported to Bio-Manguinhos, where depart periodically (according to the volume of samples) to the reference laboratory Sce Immunologie et d'Hématologie biologiques Hôpital Saint Antoine, where the dosage of antibody will be held anti epoetin alfa

SUMMARY:
The purpose of this study is to determine occurrence of pure red cell aplasia in a group of participants with chronic renal insufficiency and with resistance criteria to epoetin alfa treatment.The investigational product is producted by Bio-Manguinhos / Fiocruz (BIO-EPO) and it is provided by the Unified Health System.

ELIGIBILITY:
Inclusion Criteria:

* Use of alfa epoetin manufactured by Bio-Manguinhos for at least 8 weeks before the moment of hyporesponsiveness diagnosis;
* Nonuse of alfa epoetin from another manufacturer for at least 24 weeks before hyporesponsiveness diagnosis;
* Presence of the criteria for pure red cell aplasia disease, which is absence of a significant reduction in serum levels of leukocytes and platelets.

Exclusion Criteria:

The screened patients who have at least one of the following criteria will be excluded from the study, and it may be replaced by another participant for the research.

* if there is no legal representative, an intellectual disability that restrain the compliance and signature of informed consent,
* no agreement assigning the informed consent;
* It will be excluded from the study if from the moment of hyporesponsiveness diagnosis the participant have: lactation pregnancy, hypersensitivity or intolerance previously known for alfa epoetin or one of its components, intolerance or allergy to parenteral iron, acute hemorrhage, kidney transplantation, hemolysis defined as the presence of anemia associated with high levels of indirect bilirubin and lactate dehydrogenase , percentage of reticulocytes> 1.5% absolute reticulocyte> 75,000 / microliter.
* deficiency of folate and / or vitamin B12.
* pancytopenia.
* in use with medications known to cause anemia and / or pure red cell aplasia as: Valproic Acid; Azathioprine; Chloramphenicol; Phenytoin; Isoniazid; Mycophenolate mofetil.
* presence of the following comorbidities: Diabetes mellitus; epilepsy; chronic viral hepatitis; secondary hyperparathyroidism uncontrolled; hypertension systolic; inflammation (acute or chronic); myelofibrosis; myelodysplasia; neoplasm and thalassemias;
* severe disease in the 24 weeks before the hyporesponsiveness diagnosis; including: stroke, septic shock, thromboembolic events; acute myocardial infarction
* lack of information or damage to quality data that avoid disease classification as a case of hyporesponsiveness.
* Immunoglobulin M and Immunoglobulin M serology for Parvovirus B19, Epstein-Barr and Cytomegalovirus.
* serology for HIV in the last 12 months.
* established immunological disease.
* dosage of protein C-reactive titrated .
* presence of antinuclear antibody and rheumatoid factor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Hyporesponsiveness to EPO related to anti-alfa epoetin antibodies. | 3 years

SECONDARY OUTCOMES:
Serum levels of leukocytes and platelets correlated with anti-alfa epoetin antibodies | 3 years
Anti-alfa epoetin antibodies titers related to Hemoglobin levels | 3 years
Hemoglobin levels related to alfa epoetin dosage | 3 years
Percentage anti-alfa epoetin neutralizing antibodies related to Hemoglobin levels | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Rotman, M.D., Principal Investigator — Biomanguinhos